CLINICAL TRIAL: NCT05886101
Title: Increase Health Literacy Through Health Education Among-women Working in Readymade Garments (RMGs) to Improve Menstruation Related Self-care and Work Productivity"
Brief Title: Increase Health Literacy Through Health Education to Improve Menstruation Related Self-care and Work Productivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Rokeya Akter Bristy, Principal Investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Health literacy & productivity
Record Dates: First submitted 2023-03-29; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Work-Related Condition; Menstrual Discomfort; Occupational Problems
Keywords: Health literacy; Productivity; Menstrual self care; Health education; Occupational Nursing
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Intervention factory with health education program
  1. Health education will be provided on menstrual hygiene management and improve health literacy.
  2. Behavior change communications program
  Interventions: Behavioral: Health Education
- Control (No Intervention): No health education will be provided. However, health information material will be distributed among the participants

INTERVENTIONS:
Behavioral: Health Education — Health education will be provided to the intervention group on health literacy, self care, productivity improvement
  Arms: Intervention

SUMMARY:
The aim of the study is to increase health literacy, especially in menstruation self-care, and empower female RMG workers through health education by an occupational nurse, and as a consequent improve work productivity in RMG factories in Dhaka, Bangladesh

DETAILED DESCRIPTION:
Background: Health literacy is the degree to which an individual has the capacity to obtain, process and understand basic health information needed to make appropriate health decisions. Bangladesh is a low-income country with low health literacy levels amongst its citizens. The concept of health literacy and self-care is difficult to understand for many people. This failure to understand the concept of health literacy impacts on both the national health and the economy. Nevertheless, the health status of the garments workers is greatly affected by their working environment. Unfortunately, the factory environment is not healthy enough to protect their health. In most cases they are the main source of income in their family (Mahmud et al., 2018). Although, they are contributing in countries economy, they are suffering from different types of health problems.

Study Objective:

Increase health literacy especially in menstruation self-care and empower female RMG workers through health education by an occupational nurse, and as a consequent improve work productivity in RMG factories in Dhaka, Bangladesh

Hypothesis:

Increased health literacy amongst the women who work in RMG factories will improve the self-care practice, which consequently improves work productivity of the company.

Method: An experimental design will be used to conduct the study in RMG factories in Bangladesh. The intervention period will be for six months. A total of 4 factories are selected, which will be cluster-+randomized into the intervention group and the control group. All of them are situated in the Dhaka district. Two of them are in Mirpur Thana, one is in Ashulia upazilla, and another one is in Valuka upazilla. The intervention group will receive health education, and the control group will only receive the survey. The primary outcome is the improvement of health literacy among women working in RMGs. The secondary outcomes are improved self-care, menstrual hygiene, and empowered work productivity.

Conclusion: All interested parties would be offered the opportunity to review the results of this survey. All participants of the questionnaire would be informed of the outcomes. As the work will be carefully viewed by the student's dissertation supervisor to be of a high standard then publication in a suitable journal would be appropriate

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age (18-49 years old)
* Who is having menstruation or not
* Who will be willing to participate
* Who will like to be stay in the job for 6 months
* Who will give consent to share information for the study
* Who will willing to take part in the health educatio

Exclusion Criteria:

* Men and self-identified male or female (the third gender)

The reason: we measure menstruation practice

● Who does not belong to the assigned division or move out during the research period

(We use their data until they are present in the study)

* Who will not be willing to participate
* Who is in leave position at the time of survey

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement of health literacy measured by European health literacy scale (12-items short version) (Finbraten et al., 2018) among women in Ready Made Garments (RMG) sector in Bangladesh | 6 months
  Assessing the level of health literacy among RMG workers in Bangladesh. European health literacy scale will be used. The reporting will be done using the likert scale on a score of (1-4). Where 1 is counted as no literacy and 4 means higher literacy level. Health literacy of the garments worker will be checked by trained graduate nurses. Health education will be provided by using multimedia and data will be collected at baseline, midline and endline.

SECONDARY OUTCOMES:
Improve reproductive age women specific health literacy by using the Health literacy scale for women of reproductive age, Bangla version (From Japanese to Bangla and standardized in Study | 6 months
  Improvement on reproductive health literacy. Reproductive Women's health literacy scale. Likert scale will be used. score range is (1-4). 1= poor 2=below average, 3= good, 4 =excellent. The validity and reliability will be assessed according to the social context of Bangladesh

CONTACTS AND LOCATIONS:
Overall Officials: Michiko Moriyama, Study Chair — Hiroshima University
Locations (1):
- Rokeya Akter Bristy, Dhaka, Dhamrai, Bangladesh

IPD SHARING:
Plan to Share IPD: No